CLINICAL TRIAL: NCT03004274
Title: Running Versus Interrupted Deep Plane Sutures in Massive Weight Loss Patients: a Randomized Double Blind Study
Brief Title: Running Versus Interrupted Deep Plane Sutures in Massive Weight Loss Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Collaborators: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Principal Investigator, samer jabbour, M.D., Fondation Hôpital Saint-Joseph
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: StJo-Paris-01
Record Dates: First submitted 2016-12-18; First posted 2016-12-28 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Running sutures (Active Comparator): Deep layers will be closed using running sutures
  Interventions: Other: Running sutures
- Interrupted sutures (Experimental): Deep layers will be closed using interrupted sutures
  Interventions: Other: Interrupted sutures

INTERVENTIONS:
Other: Running sutures
  Arms: Running sutures
Other: Interrupted sutures
  Arms: Interrupted sutures

SUMMARY:
The goal of this study is to assess whether running deep wound stiches will be superior to deep interrupted stiches in body contouring surgeries in massive weight loss patients. This is a split-wound study, thereby providing an internal control within each wound. Each side of the wound will be randomized to receive one of the two suturing techniques. Patients and raters will be blinded to the suture technique used in both wound-halfs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Brachioplasty, Tighplasty, abdominoplasty, circumferential dermolipectomy in a massive weight loss patient
* The subjects are in good health
* The subject has the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator.

Exclusion Criteria:

* Under 18 years of age
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects with mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Scar cosmesis | 15 days
  The primary outcome measure of this study will be the evaluation of the scar quality. This outcome will be assessed by the Patient and Observer Scar Assessment Scale (POSAS). The patient and four blinded raters will assess the scars.
Scar cosmesis | 1.5 months
  The primary outcome measure of this study will be the evaluation of the scar quality. This outcome will be assessed by the Patient and Observer Scar Assessment Scale (POSAS). The patient and four blinded raters will assess the scars.
Scar cosmesis | 3 months
  The primary outcome measure of this study will be the evaluation of the scar quality. This outcome will be assessed by the Patient and Observer Scar Assessment Scale (POSAS). The patient and four blinded raters will assess the scars.
Scar cosmesis | 6 months
  The primary outcome measure of this study will be the evaluation of the scar quality. This outcome will be assessed by the Patient and Observer Scar Assessment Scale (POSAS). The patient and four blinded raters will assess the scars.

SECONDARY OUTCOMES:
Measurement of Scar Width | 3 months
  The width of the scar will be measured 10 centimeter from the midline on both scar-halfs.
Measurement of Scar Width | 6 months
  The width of the scar will be measured 10 centimeter from the midline on both scar-halfs.
Adverse Events | 15 days
  Noting the presence or absence of dehiscence, infection or spitting sutures.
Adverse Events | 1.5 months
  Noting the presence or absence of dehiscence, infection or spitting sutures.
Adverse Events | 3 months
  Noting the presence or absence of dehiscence, infection or spitting sutures.
Adverse Events | 6 months
  Noting the presence or absence of dehiscence, infection or spitting sutures.
Time spent suturing the wound | up to 24h
  The time spent suturing each half of the scar will be recorded in minutes
Number of suture thread needed | up to 24h
  The number of threads used to suture each half of the scar will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Josph Hospital, Paris, Paris, France